CLINICAL TRIAL: NCT03517293
Title: Enhanced Neonatal Health and Neonatal Cardiac Effect Developmentally
Acronym: ENHANCED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Carolina University (Other)
Responsible Party: Principal Investigator, Linda May, Assistant Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 12-002524
Record Dates: First submitted 2018-02-13; First posted 2018-05-07 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Physical Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: women were randomly assigned to either aerobic exercise intervention or no exercise.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of an exercise study, the participant cannot be blinded to the group. However, those assessing outcomes are blinded to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Intervention (Experimental): Aerobic Exercise training 50 minutes of moderate intensity exercise, 3 times per week from ~16-40 weeks of pregnancy
  Interventions: Behavioral: Aerobic Exercise training
- Control (No Intervention): usual daily activities - not exercise, not elevating heart rate

INTERVENTIONS:
Behavioral: Aerobic Exercise training
  Arms: Aerobic Exercise Intervention

SUMMARY:
AHA and ACSM recognize lack of exercise is a major risk factor for developing cardiovascular disease (CVD), and other CVD risk factors such as obesity. It is important to note that CVD is the sixth leading cause of death and children are more likely to be undiagnosed due to their age and lack of symptoms. Further, according to the CDC, over one-third of children and adolescents are overweight or obese and at increased risk of CVD. Although many programs for children aim to decrease CVD risks and obesity few, if any, programs begin the intervention during prenatal development. Our preliminary findings suggest that regular maternal exercise improves cardiovascular health (lower heart rate, increased heart rate variability), normalizes body fat composition, and improves nervous system and motor tone even after birth. Norepinephrine is essential for fetal development, influences many tissues (heart, nerve cells, skeletal muscle, and fat cells), and can stimulate growth factors. It is believed that exercise hormones, such as norepinephrine, released during maternal exercise influence these growth factors during development.

The central hypothesis of this proposal is that regular maternal exercise during pregnancy will improve the health of offspring before and after birth as evidenced by lower resting heart rate, increasing heart rate variability improved neurological maturation, and decreased adiposity. We have three specific aims to test this hypothesis through the Enhanced Neonatal Health and Neonatal Cardiovascular Efficiency Developmentally (ENHANCED) by Mom project (IRB approved #12-002524). Aim 1 will establish the association between maternal exercise during pregnancy and the heart health of offspring before and after birth. Aim 2 will determine the relationship between modes of regular maternal exercise and neonate neurological and muscular maturation as this relates to health of the child after birth. Aim 3 will elucidate the influence of different modes of maternal exercise during pregnancy on fetal and infant body composition as this relates to risk of obesity and CVD disease. These studies will provide novel insight into how different types of maternal exercise during pregnancy influence the overall health of offspring. Furthermore, these findings may have significant implications on the public health as it may provide evidence of pregnancy as the earliest intervention for attenuating cardiovascular disease risk of children.

DETAILED DESCRIPTION:
Recent studies have shown alarming increases in some of the major modifiable risk factors for heart disease (cholesterol, blood pressure, adiposity) in young children. We have previously found an association between self-reported exercise during pregnancy and improved heart measures of the fetus and neonate. In addition, a limited number of studies in which exercise was self-reported have demonstrated improved heart and adipose measures in the fetus or neonate with effects that persist into childhood. Previous prenatal exercise intervention studies using a prescribed exercise regimen have demonstrated the feasibility of such an approach; however, these studies have focused on maternal health and pregnancy outcomes such as birth weight. At this point, there is a gap in our understanding as to how carefully controlled, regular maternal aerobic exercise programs may lead to improvements in cardiovascular and adiposity risk factors in utero and in neonates.

The central hypothesis of this project is that maternal exercise during pregnancy will improve the health of the offspring. Specifically, the objectives of the research proposed in this application are to determine the effects of regular maternal exercise on heart function, adiposity, and neur0motor function of offspring

The data gathered will be the first documentation, by direct measurement, of the effects of maternal aerobic exercise on selected heart and obesity outcomes during the prenatal and postnatal periods. The potential impact of the proposed research on public health education regarding heart disease and obesity prevention is of public import.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 35 years BMI between 18.5 - 34.9 Pregnancy: Singleton; between 13-16 weeks gestation (based on ultrasound dating) Health Status: Healthy, no chronic illness that affects fetal growth; Clearance by Obstetric provider (no contraindications to exercise) Communication: fluent in English, available for contact by phone and email

Exclusion Criteria:

* Age: ≤ 17.9 or ≥ 35.9 years of age BMI <18.49 or >35 Pregnancy: expecting multiples; or ≥16 wks. Health Status: Any chronic condition (i.e. diabetes, hypertension, HIV, mental health disorders, etc.) that may affect fetal development Communication: unable to consent in English; No telephone/email contact Taking medicine known to affect fetal development/pregnancy outcomes (i.e. SSRI) Use of tobacco, alcohol, or other recreational drugs No transportation

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Since this is a pregnancy study, all participants are female.
Enrollment: 133 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Offspring Heart Development Measures | 36 week gestational age
  Heart Rate
Offspring Heart Development Measures | One-month after birth
  Heart Rate

SECONDARY OUTCOMES:
Offspring Adipose Development Measures | 36 week gestational age
  body fat
Offspring Adipose Development Measures | One-month after birth
  body fat
Offspring Body Development Measures | One-month after birth
  Lean Mass %

OTHER OUTCOMES:
Offspring neuromotor outomces | One-month after birth
  Neuromotor scores on PDMS-2 test

CONTACTS AND LOCATIONS:
Overall Officials: Linda E May, MS, PhD, Principal Investigator — East Carolina University
Locations (1):
- East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] May LE, McDonald S, Stewart C, Newton E, Isler C, Steed D, Sarno LA, Kelley GA, Chasan-Taber L, Kuehn D, Allman-Tucker BR, Strom C, Claiborne A, Fang X. Influence of Supervised Maternal Aerobic Exercise during Pregnancy on 1-Month-Old Neonatal Cardiac Function and Outflow: A Pilot Study. Med Sci Sports Exerc. 2023 Nov 1;55(11):1977-1984. doi: 10.1249/MSS.0000000000003227. Epub 2023 Jun 1. PMID 37259255